CLINICAL TRIAL: NCT01257334
Title: A Phase III Randomised, Double-blind, Placebo-controlled, Parallel Group, Efficacy and Safety Study of BI 10773 (10 mg, 25 mg) Administered Orally, Once Daily Over 24 Weeks in Patients With Type 2 Diabetes Mellitus With Insufficient Glycaemic Control Despite Treatment With Metformin Alone or Metformin in Combination With a Sulfonylurea
Brief Title: Patients With Type 2 Diabetes Mellitus With Insufficient Glycaemic Control Despite Treatment With Metformin Alone or Metformin in Combination With a Sulfonylurea
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Ting-I Lee, Wan Fang Hospital / Department of Metabolism
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 99050
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Experimental): BI 10773 10 mg, 25 mg administered once daily
  Interventions: Drug: BI 10773
- Control Group (Placebo Comparator): Placebo administered once daily
  Interventions: Drug: BI 10773

INTERVENTIONS:
Drug: BI 10773 — patients with type 2 diabetes mellitus with insufficient glycaemic control despite treatment with metformin alone or metformin in combination with a sulfonylurea

SUMMARY:
The objective of the current study is to investigate the efficacy, safety and tolerability of BI 10773 (10 mg, 25 mg / once daily) compared to placebo given for 24 weeks as add-on therapy to metformin or metformin plus sulfonylurea in patients with T2DM with insufficient glycaemic control.

Open-label arm: to estimate efficacy and safety of 25 mg BI 10773 in very poorly controlled patients (HbA1c > 10%)

DETAILED DESCRIPTION:
Concomitant medications, including other treatments used to treat intercurrent medical conditions during the treatment period, will be recorded on the CRFs. This record will include the name of the medication, frequency, unit dose, dosage, the date when the drug is started and stopped, and the indication for the use of the drug.

Prohibited

The following treatments are prohibited in the trial

1. Other antidiabetic agents except for the background therapy (metformin or the combination of metformin plus sulfonylurea)
2. Treatment with anti-obesity drugs or systemic steroids
3. Other investigational medications

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus prior to informed consent
* Male and female patients on a diet and exercise regimen who are pre-treated with immediate release metformin or immediate release metformin plus sulfonylurea (see below for minimum doses). The treatment regimen has to be unchanged for 12 weeks prior to randomisation.

  1. Minimum dose for metformin:

     * ≥1500 mg/day or
     * maximum tolerated dose or
     * maximum dose according to local label
  2. Minimum dose for sulfonylurea:

     * ≥half of the maximal recommended dose or
     * maximum tolerated dose or
     * maximum dose according to local label
* HbA1c of ≥ 7.0% and ≤ 10% at Visit 1 (screening) in order to be eligible for randomized treatment. HbA1c of > 10% at Visit 1 (screening) in order to be eligible for the open-label treatment arm (25 mg BI 10773)
* Age ≥ 18
* BMI ≤ 45 kg/m2 (BodyMass Index) at Visit 1 (Screening)
* Signed and dated written informed consent by date of Visit 1 in accordance with GCP and local legislation

Exclusion Criteria:

* Uncontrolled hyperglycaemia with a glucose level > 240 mg/dl (>13.3 mmol/L) after an overnight fast during placebo run-in and confirmed by a second measurement (not on the same day)
* Any other antidiabetic drug within 12 weeks prior to randomisation except those mentioned in inclusion criterion 2
* Acute coronary syndrome including myocardial infarction, stroke or TIA within 3 months prior to informed consent
* Indication of liver disease, defined by serum levels of either ALT (SGPT), AST (SGOT),or alkaline phosphatase above 3 x upper limit of normal (ULN) as determined during screening and/or run-in phase
* Impaired renal function, defined as eGFR<30 ml/min (severe renal impairment) as determined during screening and/or run-in phase
* Bariatric surgery within the past two years and other gastrointestinal surgeries that induce chronic malabsorption
* Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years
* Contraindications to metformin and/or sulfonylurea according to the local label for those patients that enter the study with the respective background therapy
* Blood dyscrasias or any disorders causing haemolysis or unstable Red Blood Cell (e.g.malaria, babesiosis, haemolytic anaemia)
* Treatment with anti-obesity drugs (e.g. sibutramine, orlistat) 3 months prior to informed consent or any other treatment at the time of screening (i.e. surgery, aggressive diet regimen, etc.) leading to unstable body weight
* Current treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent or any other uncontrolled endocrine disorder except T2D
* Pre-menopausal women (last menstruation ≤ 1 year prior to informed consent) who:

  * are nursing or pregnant or
  * are of child-bearing potential and are not practicing an acceptable method of birthcontrol, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include tubal ligation, transdermal patch, intra uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives, sexual abstinence (if acceptable by local authorities), double barrier method and vasectomised partner
* Alcohol or drug abuse within the 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures or study drug intake
* Participation in another trial with an investigational drug within 30 days prior to informed consent
* Any other clinical condition that would jeopardize patients safety while participating in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1390 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
the change from baseline in HbA1c | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ting-I Lee, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan